CLINICAL TRIAL: NCT05443139
Title: Well-being Online: Internet-based Self-administered Intervention to Reduce Anxiety and Depression Symptomatology: Randomized Clinical Trial in 7 Countries
Brief Title: Online Multi-component Psychological Intervention for Depression, Anxiety and Well-being in 7 Countries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Internacional de Valencia (Other)
Collaborators: Universidad Autonoma de Ciudad Juarez (Other); University of Guadalajara (Other); Universidad Internacional del Ecuador (Other); Universidad Santo Tomas (Other); Tilburg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Well-being_Online
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Anxiety; Depression; Wellbeing; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The Well-being Online study will implement a randomized controlled trial at five points for the intervention groups and six evaluation periods for the control group: 1)pretest, 2)middle of the treatment, 3) post-test, 4) follow up at 3 months and 5) follow up at six months. 6) Participants in the control group will be re-assigned to the intervention group after the post-waiting list period.
  The study will implement a three-arm design (parallel group), comparing:
  1. Interactive Intervention Group ,
  2. Intervention delivered through PDF files.
  3. Control group.
Who Masked: Participant
Masking Description: The patients are not aware that there are another experimental group and a control group. The conditions of the study are only known by the researcher and the Research Ethics Committee of the Universidad Autónoma de Ciudad Juárez.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive intervention (Experimental): The participants will receive a self-applied intervention composed by 10 sessions following a multi component structure. The participants assigned to this condition will count with interactive resources such as Videos, Online Forum and Exercises embedded on the platform.
  Interventions: Behavioral: Well-being online
- non-interactive intervention (Experimental): Self-administered treatment with 10 sessions will be provided through care manuals in PDF format within the same web platform. Participants in this group will receive a manual within the platform with the same content of the sessions as the experimental group but in PDF format.
  Interventions: Behavioral: Well-being online
- Waiting List group (No Intervention): The control condition consists of a 30-day waiting list, in which participants will not be able to access the interventions. After the waiting process, they will be given access to either the interactive intervention or the non-interactive intervention.

INTERVENTIONS:
Behavioral: Well-being online — Multi component Intervention composed 10 sessions following a structure based on Cognitive Behavioral Therapy (CBT), Acceptance and Commitment Therapy (ACT), Positive Psychology (PP), Mindfulness and Behavioral Activation Therapy (BAT).
  Arms: Interactive intervention; non-interactive intervention

SUMMARY:
This study evaluates the effectiveness of an online Multi-component psychological intervention, that is focused on providing self-support to the population of 5 Latin American countries and 2 European Countries. The objectives of the intervention are: 1) To reduce the symptoms of anxiety and depression in the adult population, 2) To increase the levels of subjective well-being.

DETAILED DESCRIPTION:
Anxiety and depression at clinically significant levels are associated with suicidal thoughts and behaviors. Furthermore, it is associated with the health-disease process in two ways: 1) variables that influence behavior, hindering people's healthy habits and promoting the development of unhealthy behaviors; 2) anxiety and depression affect the psycho physiological activation of people, which affects their immune system.

Considering the damage that can occur by not addressing incipient problems of anxiety and depression, it is important to develop interventions with preventive purposes. Thus, the online modality of the intervention presented in this project can benefit a significant number of people in Mexico, Ecuador, Chile, Brazil, Peru, the Netherlands and Spain. The online modality of psychological interventions is a viable treatment alternative, especially for those people who do not have any psychological treatment within their reach.

The participants will be measured at pre, middle treatment, post assessment and two follow ups of 3 and 6 months. The self-report measures will include the following Psychometrics:

1. General Anxiety Disorder with 7-items (GAD-7)
2. Center for Epidemiologic Studies Depression Scale" in its revised version (CESD-R).
3. Perceived Stress Scale (PSS-10)
4. Pittsburgh Sleep Quality scale (PSQI)
5. Action Acceptance Questionnaire II (AAQ-II)
6. The Satisfaction with Life scale
7. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS)
8. Perceived Deficits Questionnaire (PDQ-5)
9. The Positive and Negative Affect Schedule (PANAS)
10. Opinion on the treatment.
11. System usability scale.
12. Client Satisfaction Questionnaire (CSQ-8S)
13. The Telehealth Usability Questionnaire (TUQ)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Completion of 100% of the basal evaluation through the form
* Residence in one of the countries participating in the study
* Fluency/ proficiency in Spanish (Mexico, Ecuador, Chile, Peru and Spain), Dutch or English (Netherlands) or Portuguese (Brazil), depending on the country.

Exclusion Criteria:

* Participants with severe symptoms of anxiety and/or depression, or they report a diagnosis of a depression and/or an anxiety disorder.
* Participants who self-report having another diagnosed psychiatric comorbidity: personality disorder, psychotic disorder, bipolar disorder, Attention-Deficit/Hyperactivity Disorder, or others.
* Participants taking medication for symptoms of depression and/or anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Decrease in the scores of the Center for Epidemiologic Studies Depression (CESD-R) scale | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  Center for Epidemiologic Studies Depression (CES-D) is a structured self-report scale for evaluation depression symptoms. This scale assesses the number of depression symptoms within 2 weeks. The scale consists 20 items and contains 4-point score responses (0 to 3) as the following; rarely or none of the time (less than 1 day); some of a little of the time (1-2 days); occasionally or moderate amount of time (3-4 days) and most or all of the time (5-7 days). The total possible range of scores is from 0 to 60 where ^16 is the cut-off point for this scale, and higher scores indicate more symptoms of depression. It is expected a statistically significant decrease (P < 0.05) in depression symptoms.
Decrease in the score of the General Anxiety Disorder with 7-items (GAD-7) scale | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  Is a short scale with items that measure the severity of generalized anxiety disorder symptoms. Responses are based on symptoms perceived during the past week. The questions of this scale are answered in Likert format with 0-3, where the maximum total score is 21. A score between 0 and 4 points indicates that anxiety is not perceived, and a score between 15 and 21 is an indicator of perceived severe anxiety.It is expected a statistically significant decrease (P < 0.05) in anxiety symptoms.
Increase in Mental Psychological Well-being, the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Time Frame: 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  It consists of 14 items, including hedonic (i.e. affects, life satisfaction) and eudaimonic (i.e. positive relationships, psychological functioning) items, which together measure mental well-being. Each item is responded in a Likert scale (i.e. 1 = none of the time to 5 = all of the time) and the total score ranges from 14 to 70. The higher the score, the higher the mental well-being

SECONDARY OUTCOMES:
Decrease in The Perceived Stress Scale (PSS-10) | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  The PSS-10 has ten items with 5 response options (0 = Never, 1 = Almost never, 2 = Sometimes, 3 = Often, 4 = Very often). The interpretation is that the higher the score, the higher the stress level
Decrease in the score of The Pittsburgh Sleep Quality Index | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  This instrument assesses the quality patterns of sleep. It differentiates the "poor" and "good" sleep by measuring seven areas, where the range score of answers are from 0 to 3, the global sum of this scale can be a value between 0 to 60, and the cutoff point is "5" that indicates a "poor" sleep quality. It is expected a statistically significant increase (P < 0.05) in the Sleep Quality measure.
Decrease in the Action Acceptance Questionnaire II (AAQ-II) | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  The instrument measures experiential avoidance and psychological inflexibility. It consists of 7 items that are answered using a 7-point Likert scale. The items ask about the unwillingness to experience unwanted emotions and thoughts (e.g., "I am afraid of my feelings", "I worry about not being able to control my worries and feelings") and the inability to be in the present moment.
Increase in The Satisfaction with Life scale | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  It consists of 5 items in which participants must indicate how much they agree with each question, with a response option in Likert format from 1 (strongly disagree) to 7 (strongly agree). The scores range from 5 to 35, where higher scores indicate greater satisfaction with life.
Decrease in the Perceived Deficits Questionnaire or PDQ-5 | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  The scale asks about problems of functioning in daily life associated with possible cognitive problems, with a 5-point Likert-type response format, ranging from 1- Rarely to 5-Always.
Decrease negative affect in the Positive and Negative Affect Schedule (PANAS) | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  PANAS comprises two groups consisting of ten terms of either positive or negative affect. Partcipants assess their intensity on a 5-point scale ranging from "not at all" to "extremely", indicating the range of emotions at a given moment or over a period of time, and their chronic or transient nature.
Increase positive affect in the Positive and Negative Affect Schedule (PANAS) | 1 to 1.5 months, depending on the development of the patient and the completion of the 10 modules
  PANAS comprises two groups consisting of ten terms of either positive or negative affect. Partcipants assess their intensity on a 5-point scale ranging from "not at all" to "extremely", indicating the range of emotions at a given moment or over a period of time, and their chronic or transient nature.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Almela Zamorano, PhD, Study Chair — Tilburg University; Reyna Jazmín Martínez Arriaga, PhD, Study Chair — University of Guadalajara; David Villarreal Zegarra, MD, Study Chair — Instituto Peruano de Orientación Psicológica; Leivy Patricia González Ramírez, PhD, Study Chair — Tecnologico de Monterrey; Adrián Antonio Cisneros Hernández, PhD, Study Chair — University of Guadalajara; Marinna Simões Mensorio, PhD, Study Chair — Independent Researcher; Rosa Olimpia Castellanos-Vargas, PhD, Study Chair — Universidad Autónoma de Ciudad Juárez; Rogéria Lourenço dos Santos, PhD, Study Chair — Independent Researcher; Joel Omar González Cantero, PhD, Study Chair — University of Guadalajara; Viviana Sylvia Vargas Salinas, PhD, Study Chair — Independent Researcher; Joaquín Mateu Mollá, PhD, Study Chair — Universidad Internacional de Valencia; Flor Rocío Ramírez Martínez, PhD, Study Chair — Universidad Autónoma de Ciudad Juárez; Antonio Carlos Santos da Silva, MD, Study Chair — Universidad Federal da Bahia
Locations (8):
- Universidade Federal da Bahia, Ondina, Brazil
- Universidad Internacional de Ecuador, Quito, Ecuador
- Mexico (3):
  - Universidad Autónoma de Ciudad Juárez, Juárez, Chihuahua
  - Tecnólogico de Monterrey, Guadalajara
  - Universidad de Guadalajara, Guadalajara
- University of Tilburg, Tilburg, Netherlands
- Instituto Peruano de Orientación Psicológica, Lima, Peru
- Universidad Internacional de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study. The protocol of the study is currently in progress to be published, in this article will be included such study protocol, the informed consent is already shared in the register of clinical trials.
Supporting Information: ICF
Time Frame: This data will be available approximately in September 2023 and it will be permanently available. It will be shared in the databases of the journal where the article(s) will be published.
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Piqueras Rodríguez, J. A., Martínez González, A. E., Ramos Linares, V., Rivero Burón, R., García López, L. J., & Oblitas Guadalupe, L. A. (2008). Ansiedad, depresión y salud (Anxiety, depression and health). Suma Psicológica, 15, 43-74.
- [Background] Podlogar MC, Rogers ML, Stanley IH, Hom MA, Chiurliza B, Joiner TE. Anxiety, depression, and the suicidal spectrum: a latent class analysis of overlapping and distinctive features. Cogn Emot. 2018 Nov;32(7):1464-1477. doi: 10.1080/02699931.2017.1303452. Epub 2017 Mar 20. PMID 28317414
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] A-Tjak JG, Davis ML, Morina N, Powers MB, Smits JA, Emmelkamp PM. A meta-analysis of the efficacy of acceptance and commitment therapy for clinically relevant mental and physical health problems. Psychother Psychosom. 2015;84(1):30-6. doi: 10.1159/000365764. Epub 2014 Dec 24. PMID 25547522
- [Background] Bolier L, Haverman M, Westerhof GJ, Riper H, Smit F, Bohlmeijer E. Positive psychology interventions: a meta-analysis of randomized controlled studies. BMC Public Health. 2013 Feb 8;13:119. doi: 10.1186/1471-2458-13-119. PMID 23390882
- [Background] Gal E, Stefan S, Cristea IA. The efficacy of mindfulness meditation apps in enhancing users' well-being and mental health related outcomes: a meta-analysis of randomized controlled trials. J Affect Disord. 2021 Jan 15;279:131-142. doi: 10.1016/j.jad.2020.09.134. Epub 2020 Oct 7. PMID 33049431
- [Background] Ekers D, Webster L, Van Straten A, Cuijpers P, Richards D, Gilbody S. Behavioural activation for depression; an update of meta-analysis of effectiveness and sub group analysis. PLoS One. 2014 Jun 17;9(6):e100100. doi: 10.1371/journal.pone.0100100. eCollection 2014. PMID 24936656
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Carleton RN, Thibodeau MA, Teale MJ, Welch PG, Abrams MP, Robinson T, Asmundson GJ. The center for epidemiologic studies depression scale: a review with a theoretical and empirical examination of item content and factor structure. PLoS One. 2013;8(3):e58067. doi: 10.1371/journal.pone.0058067. Epub 2013 Mar 1. PMID 23469262
- [Result] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Result] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Result] Strober LB, Binder A, Nikelshpur OM, Chiaravalloti N, DeLuca J. The Perceived Deficits Questionnaire: Perception, Deficit, or Distress? Int J MS Care. 2016 Jul-Aug;18(4):183-90. doi: 10.7224/1537-2073.2015-028. PMID 27551243
- [Result] Sevilla-Gonzalez MDR, Moreno Loaeza L, Lazaro-Carrera LS, Bourguet Ramirez B, Vazquez Rodriguez A, Peralta-Pedrero ML, Almeda-Valdes P. Spanish Version of the System Usability Scale for the Assessment of Electronic Tools: Development and Validation. JMIR Hum Factors. 2020 Dec 16;7(4):e21161. doi: 10.2196/21161. PMID 33325828
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300